CLINICAL TRIAL: NCT02222935
Title: Effectiveness of Balance Training Over Routine Back Exercise in Improving Functional Outcomes of Chronic Low Back Pain Patients
Brief Title: Effectiveness of Balance Training in Chronic Low Back Pain Patients
Acronym: CLB
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskaran Chandrasekaran (Other)
Responsible Party: Sponsor-Investigator, Baskaran Chandrasekaran, Senior Physiotherapist, PSG Hospitals
Organization: PSG Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSG02
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Low Back Pain
Keywords: Balance training; low back pain; balance test; routine back exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balance exercise training (Experimental): Balance exercise training - thrice week, 2 weeks, 10 repetition Maximum/ set, 2 sets
  Interventions: Behavioral: Balance Exercise Training
- Routine Back exercise Program (Active Comparator): Routine Back exercise Program - 10 Repetition Maximum / set, 2 sets, three times weekly, 2 weeks
  Interventions: Behavioral: Routine Back exercise program

INTERVENTIONS:
Behavioral: Balance Exercise Training — Balance exercise - 5 type (single leg squat, dead lift, step ups, forward reaches), 10 Repetition Maximum, 2 sets, five times a week and 2 weeks
  Arms: Balance exercise training
Behavioral: Routine Back exercise program — Back strengthening 5 exercises - pelvic bridges, prone plank, side plank, dead bug and prone lift ups, 10 Repetition Maximum, 2 sets, five times a week, 2 weeks
  Arms: Routine Back exercise Program

SUMMARY:
Balance problems are addressed in low back pain patients. Dearth of literature available to prove core strengthening or any form of back exercises improving functional outcomes or balance in chronic back pain patients. No studies focus on balance training in improving balance of low back pain patients. The authors are conducting a randomised trial comparing balance exercises and routine back exercise program in improving pain, functional outcomes and balance of the patients

DETAILED DESCRIPTION:
Background: Balance deficits are common in low back pain. Current literature fail to prove the effectiveness of routine back exercises in improving balance of back pain patients. No study has concentrated on balance training in back pain patients.

Objective: Compare balance exercises and routine back exercises in improving balance and other functional outcomes.

Procedure: Back pain patients attending physiotherapy department of tertiary care teaching hospitals will be recruited voluntarily. Randomised to either balance and routine program based on simple lottery method. Balance training comprises of 5 exercises - single leg squats, dead lift, single leg raises, lateral step-ups and forward reach outs. Routine back exercises includes 5 sets - pelvic bridges, dynamic dead bug, prone planks, situps, lateral planks. 10Repetition Maximum, 2 Sets/ day, five days a week, 2 weeks. Baseline balance (star Edward, berg balance) and functional test (sit to stand) and pain (Visual analogue score) and post 2 weeks outcome scores will be analysed through paired and unpaired for between and within groups.

ELIGIBILITY:
Inclusion Criteria:

* non specific low back pain diagnosed by orthopedical surgeon or physiatrist
* Both genders
* Age 25 - 45 years (to avoid age related balance deficit)
* Should have balance deficit percentage (> 20%) through balance assessment scale

Exclusion Criteria:

* H/O Benign Paroxysmal Positional Vertigo
* Neuromuscular disorders(Stroke, Polio, Potts spine, spinal stenosis) affecting balance
* any form of ear infection
* Recent ear, nose, throat surgery
* Recent surgery in abdomen, thorax, head (< 2 years)
* Recent lower limb surgeries, injuries (< 6 months)
* Any form of walking aids (cane, walker)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Starr Edward Balance Test | Baseline, 2 weeks

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline, 2 weeks
Visual Analogue score | Baseline, 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pavita Devi, BPT, Principal Investigator — Senior Physiotherapist; Baskaran Chandrasekaran, MPT, Study Chair — Senior Physiotherapist; Sumathi Muraleetharan, BPT, Study Chair — Senior Physiotherpist; Ramamoorthy V Dr, MD PMR, Study Director — Head of The Department, PMR
Locations (1):
- PSG Hospitals, Department of Physical Medicine Rehabilitation, Coimbatore, Tamil Nadu, India